CLINICAL TRIAL: NCT06235580
Title: Genotype-phenotype Characterization Study on Genetic Diseases With Immune and Neurological Dysfunctions
Acronym: IFN
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMNIS2014-02
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Genetic Diseases; Immune Dysfunction; Neurological Disease; Autoimmune Diseases
MeSH Terms: conditions — Genetic Diseases, Inborn; Immune System Diseases; Nervous System Diseases; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — It is planned to use several types of samples, both fresh and frozen:
  * From blood samples, it is planned to study DNA, RNA, serum, plasma and to prepare lymphoblastic cell lines.
  * From skin samples, fibroblast cell lines will be prepared.
  * From samples of surgical waste (leftovers) of muscle and brain tissue, etc., it is planned to prepare cell cultures and search for biological markers linked to these diseases.
  * From samples of cerebrospinal fluid from surgical waste (leftovers) or from non-surgical care, it is planned to prepare cell cultures and search for biological markers linked to these diseases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients
  Interventions: Other: Biological Samples
- Controls
  Interventions: Other: Biological Samples
- Unaffected related subjects
  Interventions: Other: Biological Samples

INTERVENTIONS:
Other: Biological Samples — For patients, different types of banked frozen or fresh biological samples will be used in this research:
  * Blood
  * Skin biopsy or other tissues (liver, muscle, brain, lung...)
  * Urine
  * Saliva
  * Cerebrospinal fluid
  * Occasionally: operative "leftovers" (e.g. muscle, brain, lung tissue)
  In control patients, we would like to collect operative remnants of cell types involved in the inflammatory and/or neurological diseases studied in the laboratory, if these patients require surgery as part of their management, and if any biological material remains after surgery. Under the same conditions, a sample of cerebrospinal fluid could be recovered.
  For unaffected relatives, a single blood sample of maximum 10 ml is taken at inclusion, and samples already taken during routine care are used.

SUMMARY:
Over the past twenty years, Prof. Yanick Crow and his team have developed internationally recognized expertise in genetic pathologies affecting the immune and neurological systems. The pathologies studied have a particularly severe impact on patients' quality of life, with a high mortality rate and a significant risk of occurrence in affected families. These pathologies are rare, and very often under-diagnosed. To date, there is virtually no effective curative treatment.

Prof. Crow's team operates at the frontier between clinical and research work, and from experience, the team knows that patients and families affected by these serious pathologies are often highly motivated to help research into the pathology that affects them.

Initially, Prof. Crow's research focused primarily on the study of the genetic disease Aicardi-Goutières Syndrome (AGS). However, there is an undeniable clinical and pathological overlap between AGS and other forms of disease such as autoimmune systemic lupus erythematosus and many other genetic pathologies - e.g. familial lupus engelure, spondyloenchondromatosis and COPA syndrome. This is why research is being extended to all genetic diseases with immune and neurological dysfunctions.

DETAILED DESCRIPTION:
The research methodology is classic with regard to many genetic clinical studies, and aims to:

* clinically define the phenotypes of these diseases (in this case, genetic diseases with immune and neurological dysfunctions)
* identify the gene(s) responsible for each disease
* Understand how changes in these genes and protein functions cause these diseases.

It is possible that this research will ultimately lead to the creation of diagnostic tests (e.g. molecular diagnostic screening tests) and treatments that would be clinically very useful for the patients participating in the project. These discoveries could also improve our knowledge of other more common pathologies, particularly those associated with autoimmunity (e.g. when the body increases an immune response against its own tissues).

As a complement to this global research project, Prof. Crow's team intends to study cell populations from patients with no inflammatory pathology, in order to analyze their basal levels of immune and inflammatory mediator production, as well as to assess their capacity (kinetics and amplitude) to respond to stimuli.

ELIGIBILITY:
Inclusion criteria

* Patients :

  * Have / present a family history of genetic disease with immune and neurological dysfunction.
  * Have signed an informed consent form.
* Unaffected related subjects :

  * Be related to a patient included in this research.
  * Have signed an informed consent form.
* Control patients

  * Be free of any genetic disease with immune and neurological dysfunction.
  * Have undergone surgery as part of their management
  * Have signed an informed consent form.

Non-inclusion criteria

✓ Be deprived of liberty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be included by any hospital department involved in the management of these pathologies in France.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-12-28 (Actual); Primary Completion 2030-12-27 (Estimated); Study Completion 2035-12-27 (Estimated)

PRIMARY OUTCOMES:
Clinical features of human genetic diseases that affect the immune and neurological systems. | through study completion, an average of 1 year
  Clinical features of human genetic diseases that affect the immune and neurological systems.
Natural history of human genetic diseases that affect the immune and neurological systems. | through study completion, an average of 1 year
  Natural history of human genetic diseases that affect the immune and neurological systems.
Molecular and cellular basis of human genetic diseases that affect the immune and neurological systems. | through study completion, an average of 1 year
  Molecular and cellular basis of human genetic diseases that affect the immune and neurological systems.

CONTACTS AND LOCATIONS:
Overall Officials: Yanick Crow, MD PhD, Principal Investigator — Institut Imagine; Marie-Louise Frémond, MD, Pr, Study Chair — Institut Imagine
Locations (1):
- Necker enfants malades Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No